CLINICAL TRIAL: NCT01405105
Title: Exacerbating Factors in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Collaborators: Centocor Ortho Biotech Services, L.L.C. (Industry)
Responsible Party: Principal Investigator, Linda A Feagins, Staff Gastroenterologist, Dallas VA Medical Center
Other Study IDs: DVAMC-09-010
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with Flares of IBD: Active flare of Crohn's or UC
- Control Group: Patients with quiescent Crohn's disease or UC

SUMMARY:
Cross-sectional study of potential triggers for flares of Crohn's disease or ulcerative colitis.

DETAILED DESCRIPTION:
Detailed questionnaires with patient in regards to potential triggers for flares of IBD. Includes both patients with flares and those in remission as a control group.

ELIGIBILITY:
Inclusion Criteria:

* History of verified Crohn's disease or ulcerative colitis

Exclusion Criteria:

* unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Flare of Crohn's disease Flare of ulcerative colitis Quiescent IBD (control)
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2009-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Frequency of identifiable trigger for flare | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Feagins, MD, Principal Investigator — Dallas VA Medical Center
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States